CLINICAL TRIAL: NCT05443516
Title: Disease Activity Biomarkers in Patients With Systemic Lupus Erythematosus. Recherche de Biomarqueurs de l'activité de la Maladie Chez Des Patients Atteints de Lupus érythémateux disséminé.
Brief Title: Disease Activity Biomarkers in Patients With Systemic Lupus Erythematosus
Acronym: JD001
Status: Recruiting | Type: Observational
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Sponsor
Other Study IDs: 2014/07AVR/170
Record Dates: First submitted 2022-06-17; First posted 2022-07-05 (Actual); Last update posted 2022-07-05 (Actual); Status verified 2022-06

CONDITIONS: Lupus Nephritis
MeSH Terms: conditions — Lupus Nephritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — residual blood and urine
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Systemic Lupus Erythematosus - Lupus Nephritis Cohort: Systemic Lupus Erythematosus - Lupus Nephritis Cohort

SUMMARY:
The aim of this research project is to better understand the origin and clinical significance of two lupus-specific "genetic signatures" (IFN signature and plasma cell signature) in patient subgroups with well-defined clinical characteristics. Our aim is to correlate these genetic signatures with cell activation profiles and the production of specific cytokines in different populations from whole blood and in short-term cultures of these circulating cells.

DETAILED DESCRIPTION:
The aim of the experiment is, on the one hand, to identify and study the different cell populations from whole blood by flow cytometry and, on the other hand, to assay different cytokines in blood and urine samples from diseased (SLE) and control subjects (with non-inflammatory rheumatic diseases) in order to highlight and correlate the presence of biomarkers to disease activity or to a clinical manifestation of the disease.

In vitro studies will also be carried out on short-term cultures of PBMCs (Peripheral Blood Mononuclear Cells).

ELIGIBILITY:
Inclusion Criteria:

* Fulfilment of the EULAR/ACR classification criteria of SLE.
* 18 years of age or above.
* Incident or Flare biopsy-proven proliferative or membranous LN

Exclusion Criteria:

* Antiphospholipid syndrome nephropathy (APSN).
* Pregnancy at baseline (pregnancy during follow-up will not lead to exclusion).
* Anticipated non-adherence to therapy.
* Medical conditions interfering with outcome evaluations.
* Inability to read and/or sign the informed consent form.

Ages: 18 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Incident or Flare biopsy-proven proliferative or membranous LN diagnosis
Sampling Method: Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2014-06-16 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2032-12-31 (Estimated)

PRIMARY OUTCOMES:
Biomarker analysis of lupus nephritis activity - whole blood cell populations | baseline
  whole blood cell populations - flow cytometry assay
Biomarker analysis of lupus nephritis activity - blood cytokines | baseline
  blood cytokines - flow cytometry assay
Biomarker analysis of lupus nephritis activity - urine cytokines | baseline
  urine cytokines - flow cytometry assay

CONTACTS AND LOCATIONS:
Overall Officials: Frédéric Houssiau, Pr, Principal Investigator — Cliniques universitaires Saint-Luc- Université Catholique de Louvain
Locations (1):
- Cliniques universitaires Saint-Luc, Brussels, Belgium